CLINICAL TRIAL: NCT01338571
Title: The Effect of Resistant Starch on the Stool Microflora of Children: A Pilot Study
Brief Title: Horton & Maizy Pilot Study for Resistant to Starch
Status: Completed | Type: Observational
Sponsor: Pennington Biomedical Research Center (Other)
Responsible Party: Principal Investigator, Frank Greenway, Principal Investigator, Pennington Biomedical Research Center
Other Study IDs: PBRC 28012
Record Dates: First submitted 2011-04-15; First posted 2011-04-19 (Estimated); Last update posted 2015-12-18 (Estimated); Status verified 2015-12

CONDITIONS: pH; Weight Gain
Keywords: stool fatty acid
MeSH Terms: conditions — Weight Gain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: None Retained — collect 3 daily stool samples are retained at baseline and after 4 weeks
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Healthly children: Children will be given yogurt twice a day for four weeks. The dose for an adult is 8 ounces of yogurt twice a day. The dose will be scaled to the children based upon surface area dosing charts, but will not exceed a resistant starch load of 1 gram per year of age plus 10 grams10.

SUMMARY:
This is a pilot study and will be used to power an NIH grant application on the effect of resistant starch on weight gain in children.

DETAILED DESCRIPTION:
Stool fatty acids and stool pH from the baseline and week 4 stool samples will be compared by paired-t test. The stool microflora changes will be reported using descriptive statistics for the percent changes in the different bacterial phyla.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female between the ages of 5 and 15 years

Exclusion Criteria:

* Gastrointestinal disease
* Medication such as antibiotics that have the potential for altering the gut bacterial flora.
* Allergic to milk or corn products.

Ages: 5 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children between ages 5 and 15
Sampling Method: Probability Sample
Enrollment: 4 (Actual)
Dates: Start 2008-02; Primary Completion 2008-05 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Effect of resistant starch on weight gain in children | Four weeks
  During the 4 weeks while still consuming the yogurt supplements, 3 daily stool samples will be collected in the same manner as the baseline stool collections. Stool fatty acids from the baseline and week 4 stool samples will be compared by paired-t test. The stool microflora changes will be reported using descriptive statistics for the percent changes in the different bacterial phyla.

SECONDARY OUTCOMES:
Effect of resistant starch on weight gain in children | Four weeks
  During the 4 weeks while still consuming the yogurt supplements, 3 daily stool samples will be collected in the same manner as the baseline stool collections. Stool pH from the baseline and week 4 stool samples will be compared by paired-t test. The stool microflora changes will be reported using descriptive statistics for the percent changes in the different bacterial phyla.

CONTACTS AND LOCATIONS:
Locations (1):
- Pennington Biomedical Research Center, Baton Rouge, Louisiana, United States